CLINICAL TRIAL: NCT05728892
Title: Melatonin and Its Effect on the Perioperative Opioid Needs in Pediatric Patients Undergoing Laparoscopic Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAMSU R264/2022
Record Dates: First submitted 2023-01-26; First posted 2023-02-15 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): patients undergoing abdominal surgery receiving melatonin
  Interventions: Drug: Melatonin 3 MG
- Group B (Placebo Comparator): control group
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin 3 MG — Preopertive melatonin adminstration oral 0.2 mg /kg 45 min before general anaethesia.
  Arms: Group A
Other: Placebo — Placebo medication will be given to control group
  Arms: Group B

SUMMARY:
To study the role of Preoperative Melatonin adminsteration in pediatric patients undergoing laparoscopic surgeries regarding its analgesic and sedative effects

ELIGIBILITY:
Inclusion Criteria:

* Age from 2 to 10 years.
* Sex: Both sexes.
* Patients with ASA classificaion I and II.

Exclusion Criteria:

* Declining to give written informed consent.
* History of allergy to the medications used in the study.
* psychiatric disorder.
* ASA classification III-V.
* Fever ,cough , asthma or upper respiratory tract infection, neuromuscular disorders, spine abnormalities.
* Anticipated difficult airway .
* History of malignant hyperthermia

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Discharge from postanesthesia care unit (1 hour)
  Assesment of pain will be done using Face, Leg, Activity , Crying and Consolability behavioural pain scale (FLACC), Each category is scored on the 0-2 scale, which results in a total score of 0-10.
  0 = Relaxed and comfortable, 1-3 = Mild discomfort, 4-6 = Moderate pain and 7-10 = Severe discomfort or pain or both.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university hospital, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No